CLINICAL TRIAL: NCT06778863
Title: GUARDIAN-101: A Phase 1 Dose Escalation and Expansion Study of CLSP-1025 in Adult Patients With Solid Tumors That Harbor the p53 R175H Mutation
Brief Title: A Study of CLSP-1025 in Adult Patients With Solid Tumors That Harbor the p53 R175H Mutation
Acronym: GUARDIAN-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Clasp Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLSP-1025-101
Record Dates: First submitted 2025-01-08; First posted 2025-01-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Unresectable Solid Tumor; Metastatic Solid Tumor; Colorectal Adenocarcinoma; Pancreatic Adenocarcinoma; Lung Cancer; Ovarian Cancer; Breast Cancer; Head and Neck Squamous Cell Carcinoma; Prostate Cancer; Bladder Cancer
Keywords: CLSP-1025; T Cell Engager; TCE; TP53
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Monotherapy Dose Escalation of CLSP-1025 (Experimental): Dose escalation of CLSP-1025 in HLA-A*02:01-positive adult patients with advanced solid tumors that harbor the p53 R175H mutation
  Interventions: Drug: CLSP-1025
- Part B: Monotherapy Dose Expansion of CLSP-1025 (Experimental): Dose expansion of CLSP-1025 in HLA-A*02:01-positive adult patients with advanced solid tumors that harbor the p53 R175H mutation
  Interventions: Drug: CLSP-1025

INTERVENTIONS:
Drug: CLSP-1025 — CLSP-1025 will be administered by IV infusion

SUMMARY:
Phase 1 dose escalation and expansion study of CLSP-1025, a first-in-class HLA-A*02:01 specific T cell engager (TCE) targeting solid tumors that harbor the p53 R175H mutation.

DETAILED DESCRIPTION:
This Phase 1, open-label, multicenter study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of CLSP-1025 when administered to HLA-A*02:01-positive adult patients with advanced solid tumors that harbor the p53 R175H mutation. The study will be conducted in 2 parts: Part A Monotherapy Dose Escalation to determine the recommended dose(s) for expansion (RDE[s]) and Part B Monotherapy Expansion to explore the preliminary antitumor activity as well as further characterize the safety, tolerability, PK, and PD of CLSP-1025 at the RDE(s).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be at least 18 years of age at the time of signing the informed consent.
* Patients must be willing and able to provide written informed consent
* Patients must have locally advanced or metastatic solid tumors that have progressed after standard of care therapy or for which no standard therapy exists
* Tumors must harbor a TP53 R175H variant mutation confirmed by an accredited laboratory-based test
* Patients must be HLA-A*02:01 positive by central assay
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at the time of enrollment
* Adequate hematological, renal and hepatic function
* Per Investigator judgement, patient is willing and able to complete study visits and/or procedures per the protocol and comply with study requirements for study participation

Key Exclusion Criteria:

* Patients with Li-Fraumeni syndrome or other known germline p53 R175H mutation
* Patients who have received other p53 R175H-directed therapies
* Patients who have not fully recovered from adverse events due to previous anticancer therapies
* Patients with active infection requiring systemic antimicrobial therapy
* Any other primary malignancy within the 2 years prior to enrollment (except for non- melanoma skin cancer, carcinoma in situ (eg, cervix, bladder, breast) or prostate cancer in remission.
* Known active central nervous system metastases and/or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Part A: Determine the maximum tolerated dose (MTD) and/or the recommended dose(s) for expansion (RDE[s]) | 28 days after infusion
  Rate of dose-limiting toxicities (DLTs) after infusion of CLSP-1025
Part B: Evaluate the Objective response rate (ORR) of CLSP-1025 as a monotherapy in HLA-selected patients with advanced solid tumors that express the p53 R175H mutation | Up to 24 months after infusion
  Objective response rate (ORR) per RECIST V1.1 determined by Investigator assessment

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events, as assessed by CTCAE, v5.0 | Up to 24 months after infusion
  Incidence and severity of treatment-emergent adverse events (TEAEs)
Number of patients with treatment-related adverse events, as assessed by CTCAE, v5.0 | Up to 24 months after infusion
  Incidence and severity of treatment-related adverse events (TRAEs)
Number of patients with clinically significant changes in QTcF Interval | Up to 24 months after infusion
  Incidence of clinically significant changes in QTcF Interval
Maximum plasma concentration (Cmax) of CLSP-1025 | Pre-dose and up to 168 hours post-dose
  To determine the maximum plasma concentration (Cmax) of CLSP-1025
Minimum plasma concentration (Cmin) of CLSP-1025 | Pre-dose and up to 168 hours post-dose
  To determine the minimum plasma concentration (Cmin) of CLSP-1025
Area under the curve at the end of the dosing interval (AUCtau) of CLSP-1025 | Pre-dose and up to 168 hours post-dose
  To determine the area under the curve at the end of the dosing interval (AUCtau) of CLSP-1025
Half-life (t1/2) of CLSP-1025 | Pre-dose and up to 168 hours post-dose
  To determine the half-life (t1/2) of CLSP-1025
Assess the immunogenicity of CLSP-1025 | Up to 24 months after infusion
  To determine the presence of anti-CLSP-1025 antibodies at baseline and on treatment
Part A: Objective Response Rate (ORR) | Up to 24 months after infusion
  Determine Objective Response Rate (ORR) per RECIST V1.1
Duration of response (DOR) | Up to 24 months after infusion
  Determine DOR of CLSP-1025 until radiographic disease progression per RECIST V1.1 or death
Time to Response | Up to 24 months after infusion
  Determine time to response of CLSP-1025 per RECIST V1.1.
Disease Control Rate | Up to 24 months after infusion
  Determine disease control rate of CLSP-1025 per RECIST V1.1.
Progression-free survival (PFS) | Up to 24 months after infusion
  Determine PFS of CLSP-1025 until radiographic disease progression per RECIST V1.1 or death.
Time of Treatment | Up to 24 months after infusion
  Determine Time on Treatment of CLSP-1025 from first dose to last dose
Overall Survival (OS) | Up to 24 months after infusion
  Determine OS of CLSP-1025 until death

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - USC - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - The University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute (SCRI) Oncology Partners, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No